CLINICAL TRIAL: NCT04960969
Title: The Effects of Time-Restricted Eating Model on Eating Behaviors, Impulsivity and Food Intake
Brief Title: The Effects of Time-Restricted Eating Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elif Emiroğlu (Other)
Responsible Party: Sponsor-Investigator, Elif Emiroğlu, Lecturer, Istinye University
Organization: Istinye University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TRF
Record Dates: First submitted 2021-07-09; First posted 2021-07-14 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Time Restricted Feeding; Feeding Behavior; Impulsive Behavior
MeSH Terms: conditions — Intermittent Fasting; Feeding Behavior; Impulsive Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted Feeding Group (Experimental): Participants will apply time-restricted feeding (8 hours/day) for 28 days.
  Interventions: Other: Time-restricted feeding for 4 weeks
- Control Group (No Intervention): No intervention will be applied.

INTERVENTIONS:
Other: Time-restricted feeding for 4 weeks — Participants in this group will follow a time-restricted diet for 28 days. Consumption of only non-energy drinks will be allowed for 16 hours. During the 8-hour eating period, there will be no restriction on the content of the diets.
  Arms: Time-restricted Feeding Group

SUMMARY:
There is increasing evidence of the effects of the time-restricted diet model based on the daily intake of energy within a period of 8-12 hours on body weight control and metabolic parameters. There is no study on the potential effects of this nutritional model, which is thought to be an effective strategy in struggling with metabolic syndrome, on individuals' eating behavior and impulsivity levels. This study, which aims to evaluate the effects of time- restricted diet strategy on food intake, eating attitude and behavior and impulsivity level in adults, is a mixed method, randomized controlled intervention study. Thirty adult individuals between the ages of 18-65 will be included in this study, which will be carried out between 31.05.2021-31.12.2021 in Istinye University. Participants will be divided into 2 groups: the intervention group (n = 15) will apply a time-restricted nutrition model for 4 weeks, and no intervention will be applied to the control group (n = 15). Participants' food intake before and after the intervention period will be evaluated with a 3-day food intake record, their eating attitudes will be evaluated with the Eating Attitude Test (EAT-26), their impulsivity levels will be evaluated with the Barratt Impulsiveness Scale-Short Form (BIS-11-SF) and Go / NoGo test, and their eating behaviors will be evaluated with the Three Factor Eating Questionnaire (TFEQ-R21). At the end of the research, all individuals in the intervention group will be interviewed in depth and their experiences regarding the process will be recorded. IBM SPSS 22 program will be used in the analysis of all quantitative data, and the MAXQDA-12 program will be used in the analysis of qualitative data. The data obtained from this research will clear up the applicability of the time- restricted diet model and its effects on eating behaviors of adults.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Body mass index (BMI) ≥ 18.5 kg/m2,
* Routine eating window ≥10 hours (including all energy-containing meals and drinks),
* To agree to participate in the research voluntarily.

Exclusion Criteria:

* Age <18 or >65,
* BMI <18.5 kg/m2,
* To have applied nutritional therapy for weight loss or medical treatment in the last 6 months,
* Being in pregnancy or lactation period,
* Working the night shift or the partner working the night shift (if it affects the participant's sleep and nutritional status),
* Having a known neurological or psychological disorder,
* Declaring that have a history of eating disorder in the last 3 months,
* Weight change of ≥ 5 kg in the last 3 months,
* Having an uncontrolled medical problem (cardiovascular, pulmonary, rheumatological, hematological, oncological, gastrointestinal, psychiatric, endocrinological, etc.)
* Receiving medical treatment that may have a significant impact on glucose metabolism, appetite or energy balance,
* Being on antidepressant treatment,
* Having a history of bariatric surgery,
* Having celiac, crohn's or ulcerative colitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in food intake of participants | Baseline and Week 4
  The food intake of the participants will be determined by the 3-day food consumption record at the beginning and at the 4th week.
Changes in impulsivity level of participants | Baseline and Week 4
  The impulsivity of the participants will be determined by the Go/NoGo Task and Short form of Barratt Impulsiveness Scale (BIS-11-SF) at the beginning and at the 4th week.
Changes in eating attitude of participants | Baseline and Week 4
  The eating attitude of the participants will be determined by the Eating Attitude Test (EAT-26) at the beginning and at the 4th week.
Changes in eating behaviors of participants | Baseline and Week 4
  The eating behaviors of the participants will be determined by the Three Factor Eating Questionnaire (TFEQ-R21) at the beginning and at the 4th week.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adafer R, Messaadi W, Meddahi M, Patey A, Haderbache A, Bayen S, Messaadi N. Food Timing, Circadian Rhythm and Chrononutrition: A Systematic Review of Time-Restricted Eating's Effects on Human Health. Nutrients. 2020 Dec 8;12(12):3770. doi: 10.3390/nu12123770. PMID 33302500
- [Background] Flanagan A, Bechtold DA, Pot GK, Johnston JD. Chrono-nutrition: From molecular and neuronal mechanisms to human epidemiology and timed feeding patterns. J Neurochem. 2021 Apr;157(1):53-72. doi: 10.1111/jnc.15246. Epub 2020 Dec 10. PMID 33222161
- [Background] Quist JS, Jensen MM, Clemmensen KKB, Pedersen H, Bjerre N, Storling J, Blond MB, Wewer Albrechtsen NJ, Holst JJ, Torekov SS, Vistisen D, Jorgensen ME, Panda S, Brock C, Finlayson G, Faerch K. Protocol for a single-centre, parallel-group, randomised, controlled, superiority trial on the effects of time-restricted eating on body weight, behaviour and metabolism in individuals at high risk of type 2 diabetes: the REStricted Eating Time (RESET) study. BMJ Open. 2020 Aug 26;10(8):e037166. doi: 10.1136/bmjopen-2020-037166. PMID 32847912
- [Background] Moon S, Kang J, Kim SH, Chung HS, Kim YJ, Yu JM, Cho ST, Oh CM, Kim T. Beneficial Effects of Time-Restricted Eating on Metabolic Diseases: A Systemic Review and Meta-Analysis. Nutrients. 2020 Apr 29;12(5):1267. doi: 10.3390/nu12051267. PMID 32365676
- [Background] Pellegrini M, Cioffi I, Evangelista A, Ponzo V, Goitre I, Ciccone G, Ghigo E, Bo S. Effects of time-restricted feeding on body weight and metabolism. A systematic review and meta-analysis. Rev Endocr Metab Disord. 2020 Mar;21(1):17-33. doi: 10.1007/s11154-019-09524-w. PMID 31808043
- [Background] Regmi P, Heilbronn LK. Time-Restricted Eating: Benefits, Mechanisms, and Challenges in Translation. iScience. 2020 Jun 26;23(6):101161. doi: 10.1016/j.isci.2020.101161. Epub 2020 May 15. PMID 32480126
- [Derived] Guner E, Aktac S. Time-restricted feeding can increase food-related impulsivity: a randomized controlled trial. Nutr Neurosci. 2025 Jan;28(1):28-36. doi: 10.1080/1028415X.2024.2344139. Epub 2024 Apr 22. PMID 38648081